CLINICAL TRIAL: NCT00003261
Title: Treatment of HIV-Related Primary Central Nervous System Lymphoma (HIV-PCNSL): A Phase II Trial With Neoadjuvant Chemotherapy (High-Dose Methotrexate (MTX) Plus High-Dose Zidovudine) and Radiotherapy
Brief Title: Chemotherapy and Radiation Therapy in Treating Patients With HIV-Related Primary Central Nervous System Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centro di Riferimento Oncologico - Aviano (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000066153; ITA-GICAT-POS1; EU-97018
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2001-10

CONDITIONS: Lymphoma
Keywords: AIDS-related primary CNS lymphoma
MeSH Terms: conditions — Lymphoma | interventions — Methotrexate; Zidovudine; Neoadjuvant Therapy; Radiotherapy

INTERVENTIONS:
Drug: methotrexate
Drug: zidovudine
Procedure: neoadjuvant therapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining radiation therapy with chemotherapy may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving methotrexate and zidovudine together with radiation therapy works in treating patients with HIV-related primary central nervous system lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of neoadjuvant chemotherapy and radiation therapy in the treatment of HIV-related primary CNS lymphoma patients.
* Evaluate the toxicity and overall survival of these patients.

OUTLINE: Patients receive chemotherapy consisting of high-dose methotrexate IV administered on day 1 and high-dose zidovudine IV administered on days 1-3 every 2 weeks. Patients receive 3 courses of therapy. Following chemotherapy, patients receive radiation therapy to the lesion site daily.

Patients are followed every 3 months for 1 year and then every 6 months thereafter.

PROJECTED ACCRUAL: This study will accrue 14 patients.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven HIV-related non-Hodgkin's lymphoma of the CNS
* No systemic lymphoma

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* WHO 0-3

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 3000/mm^3
* Platelet count at least 80,000/mm^3

Hepatic:

* No serious impairment of liver function

Renal:

* No serious impairment of renal function
* Creatinine clearance at least 40 mL/min

Cardiovascular:

* No serious impairment of cardiac function

Neurologic:

* Neurological functional status 0-3

Other:

* No prior or active CNS-opportunistic infections
* No AIDS dementia complex
* No active systemic infections

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy or radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 1997-05

PRIMARY OUTCOMES:
Efficacy
Toxicity
Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Umberto Tirelli, MD, Study Chair — Centro di Riferimento Oncologico - Aviano
Locations (1):
- Centro di Riferimento Oncologico - Aviano, Aviano, Italy